CLINICAL TRIAL: NCT04485533
Title: Clinical Investigation to Assess the Efficacy and the Safety of VisuXL® Ophthalmic Gel Administered in Patients Affected by Moderate Dry Eye Disease (DED): a Randomized, Cross Over, Double Blind Study
Brief Title: Clinical Investigation to Assess the Efficacy and the Safety of VisuXL® Gel Administered in Patients Affected by Moderate DED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VF-OS-004/2019
Record Dates: First submitted 2020-06-02; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VisuXL® Gel/HYLO® (Experimental): Patients treated with VisuXL® ophthalmic gel for the first 30 days (1 treatment period) and with HYLO® for the second 30 days (2 treatment period).
  Interventions: Device: VisuXL® Gel; Device: HYLO®
- HYLO®/VisuXL® Gel (Active Comparator): Patients treated with HYLO® for the first 30 days (1 treatment period) and with VisuXL® ophthalmic gel for the second 30 days (2 treatment period).
  Interventions: Device: VisuXL® Gel; Device: HYLO®

INTERVENTIONS:
Device: VisuXL® Gel — VisuXL® ophthalmic gel, available in a multidose 10ml bottle without preservatives based on Coenzyme Q10, Vitamin E TPGS and cross-linked sodium carboxymethylcellulose.
  Dose/dosage: 1 drop per eye twice a day.
Device: HYLO® — HYLO® ophthalmic solution, a phosphate- and preservative-free sterile eye drops containing 2 mg/ml of hyaluronic acid sodium salt, a citrate buffer, sorbitol and water.
  Dose/dosage: 1 drop per eye twice a day

SUMMARY:
This is a post-market, european multicenter study. This is a randomized, cross-over, double blind study with competitive enrolment, aimed to enroll a total of 90 patients with a diagnosis of moderate dry eye disease (DED).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the non-inferiority of the new treatment versus the comparator.

Patients, after signing the Informed Consent, will enter into a 1-week screening phase during which the baseline tests will be conducted.

Baseline (V0), Day 30 ± 1 week (V1), Day 38 ± 2 days (V2), Day 68 ±1 week (V3) of treatment.

Between V1 and V2 one week of wash out should be performed. Of note, all ophthalmologic evaluations listed in the Flow-Chart will be performed on both eyes of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed.
* Males and Females aged ≥18 years at the time of the signature of ICF.
* Patients with moderate dry eye disease (DED) according to IDEEL questionnaire (score ≥51 and ≤64) and diagnosed at least 3 months before enrolment.
* No use of other tear substitutes in the 5 days prior to enrolment, except for refresh solutions.
* TBUT value <6 sec.
* Willing to follow all study procedures, including attending all site visits, tests and examinations.
* Women must agree to be using two forms of effective contraception, be post-menopausal from at least 12 months prior to trial entry, or surgically sterile.

Exclusion Criteria:

* Patients with a mild or severe dry eye disease (DED) according to IDEEL questionnaire (score ≤50 and ≥65, respectively).
* Use of ophthalmologic products in the 14 days prior to enrolment, except for refresh solutions and stable glaucoma treatment.
* No previous history or presence of any disease involving cornea or conjunctiva.
* Sjӧgren syndrome.
* History or active cicatricial conjunctivitis.
* History of ocular surface burns.
* Use of contact lenses.
* Corneal refractive surgery 1 year post-operative.
* Any ocular surgery in the previous 3 months preceding the study.
* Unstable glaucoma (treatment changes in the last year).
* Any macular or retinal disease that could impact visual acuity.
* Best corrected visual acuity (BCVA) below 20/40.
* Blepharitis treatment started less than 3 months before enrolment.
* Neurological, neurodegenerative or cerebrovascular conditions.
* Any clinically significant history of serious digestive tract, liver, kidney, cardiovascular, cancer or hematological disease.
* Unstable treatment with systemic medications, such as diuretics, antihistamines, antidepressants, psychotropics, cholesterol lowering agents and beta-blockers.
* Known hypersensitivity to one of the administered products.
* Known drug and/or alcohol abuse.
* Mental incapacity that precludes adequate understanding or cooperation.
* Participation in another investigational study or blood donation within 1 month prior to ICF signature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Tear Break-Up Time (TBUT) | through study completion, an average of 2.5 months
  To evaluate the effect of treatment with VisuXL® GEL versus HYLO® on the stability of the tear film by Tear Break-Up Time (TBUT) in patients affected by moderate dry eye disease (DED).

SECONDARY OUTCOMES:
Stability of the tear film assessed by NIBUT (Non-invasive Break-Up Time) | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Stability of the tear film
Functional Visual Acuity (FVA) | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Functional Visual Acuity (FVA)
Tear secretion | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Tear secretion
Burning, foreign body sensation, itching, and photophobia symptoms of DED assessed by Visual Analogue Scale (10 points VAS) | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Burning, foreign body sensation, itching, and photophobia symptoms of DED.
  (VAS: scale where patient has to specify level of satisfaction by indicating a position along a continuous line between two end-points (0 - 10). 0 indicates no satisfaction while 10 represents the highest level).
Conjunctival inflammation assessed by staining grade with Van Bijsterveld Scale | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Conjunctival and corneal inflammation
Corneal inflammation assessed by staining grade with SICCA Scale | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Conjunctival and corneal inflammation
Impact of DED on Everyday Life assessed by means of Quality of Life questionnaire IDEEL | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Impact of DED on Everyday Life assessed by means of Quality of Life questionnaire IDEEL
Each of the three modules that are part of IDEEL questionnaire | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Each of the three modules that are part of IDEEL questionnaire
Number of participants with treatment-related Adverse Events and Adverse Device Events assessed in a descriptive way | through study completion, an average of 2.5 months
  To evaluate the time-related effects of treatment with VisuXL® GEL versus HYLO® in patients affected by moderate dry eye disease (DED) on Medical devices' safety and tolerability:
  * Allergy to any device compound
  * Any other adverse event (AE)
  * Adverse device effects (ADEs) -Undetected/unforeseen manufacturing ADE which might bring to application procedure errors -
  * Contamination of the device nozzle and possibility to contaminate both eyes
  * Interaction with any other permitted local administered therapy
  * Vital signs: blood pressure (BP), heart rate (HR), respiratory rate (RR)

CONTACTS AND LOCATIONS:
Locations (3):
- Hôpital Morvan, Brest, Finistère, France
- ASST-Santi Paolo e Carlo-Presidio San Paolo, Milan, MI, Italy
- Hospital Clínico San Carlos de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No